CLINICAL TRIAL: NCT06969755
Title: Biomarkers to Enhance Early Schizophrenia Treatment
Acronym: BEEST
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BEEST; 1R01MH134883-01A1 (NIH)
Record Dates: First submitted 2025-04-04; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Schizophenia Disorder
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole; Risperidone; Clozapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- risperidone (Active Comparator): risperidone treatment provided per protocol
  Interventions: Drug: risperidone
- aripiprazole (Active Comparator): aripiprazole treatment per protocol
  Interventions: Drug: aripiprazole
- clozapine (Active Comparator): clozapine treatment per protocol
  Interventions: Drug: clozapine

INTERVENTIONS:
Drug: aripiprazole — aripiprazole arm (titrated dose)
  Arms: aripiprazole
Drug: risperidone — risperidone arm (titrated dose)
  Arms: risperidone
Drug: clozapine — clozapine (titrated dose)
  Arms: clozapine

SUMMARY:
This study is recruiting participants who are experiencing a first episode of psychosis and who have certain genetic factors that may make them respond better to certain medications that are used to treat people with psychosis.

DETAILED DESCRIPTION:
The study is designed to test the hypothesis that, compared with standard treatment with FL-APs (risperidone or aripiprazole), early treatment with clozapine (CLZ) will benefit patients in the first episode of psychosis (FEP) who have been designated three biomarker positive (3B+) as follows: 1) likely to have a poor response to FL-APs; 2) not at heightened risk for clozapine-induced agranulocytosis and 3) not at heightened risk for antipsychotic-induced weight gain. The study will recruit n=410 FEP across the 5 participating sites for screening on each of the 3 biomarkers (striatal connectivity in relation to risk of treatment response/resistance to conventional antipsychotics, MC4R genotype in relation to weight gain risk, and HLA-DQB1 genotype in relation to agranulocytosis risk), which involves a rs-fMRI scan (for response/non-response prediction) and a blood draw for genotyping per above (to screen for heightened risk for each of the two side effects). Those failing to meet any of the 3 biomarker criteria will receive FEP care but will not be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 35.
2. DSM5 diagnosis (as determined by the SCID5) of schizophrenia, schizoaffective disorder, schizophreniform disorder.
3. Current positive symptoms rated ≥4 (moderate) on one or more of the following BPRS positive subscale items: unusual thought content, conceptual disorganization, hallucinatory behavior, suspiciousness.
4. Preserved striatal connectivity, as determined by screening MRI scan
5. Absence of the MC4R high-risk genotype, as determined by genetic testing
6. Absence of the HLA-DQB1 high-risk genotype, as determined by genetic testing
7. In an early phase of illness as defined by having taken antipsychotic drugs for a cumulative lifetime period of 4 weeks or less (with exceptions of very low doses for other off-label indications, e.g. sleep)
8. Ability to provide informed consent

Exclusion Criteria:

1. The patient reports or medical records state a serious neurological or endocrine disorder at screening that the investigator determines could interfere with the interpretation of the efficacy or safety measurements
2. An abnormal EKG at screening that the investigator determines could interfere with the interpretation of the efficacy or safety measurements
3. Any medical condition which requires treatment with a medication with psychotropic effects.
4. Significant risk of suicidal or homicidal behavior (i.e. 'severe' risk on the Columbia Suicide Scale, a 'hostility' score of 7 on the BPRS, or an answer of 'yes' on questions 4,5 or 6 on the CDSS).
5. Cognitive limitations, or any other factor that would preclude potential participants providing informed consent
6. Contraindications to MRI (e.g. pacemaker).
7. Meeting SCID-5 substance use disorder moderate or severe for any substance, other than nicotine within 3 months of screening visit. Meeting SCID5 substance use disorder mild for any substance other than cannabis, alcohol, or nicotine for less than 3 months prior to screening visit, or a positive urine baseline drug screen with a substance other than nicotine, alcohol, or cannabis
8. Suspected DSM5 intellectual disability based upon clinical interview and psychosocial history, as well as screening with the Weschler Test for Adult Reading (IQ score <71)
9. Prior psychosurgery
10. Pregnancy (self-report)
11. Seizure disorder (self-report)

    -

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2030-07-30 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
Total change in BPRS Symptoms | 12 weeks
  To compare the 12-week response rate of CLZ versus FL-APs (both risperidone and aripiprazole) utilizing the BPRS

SECONDARY OUTCOMES:
Weight Gain | 12 weeks
  To compare weight gain associated with 12 weeks of treatment with CLZ vs. FL-APs in 3B+ FEP patients.
Agranulocytosis | 12 weeks
  To compare rates of agranulocytosis in 3B+ FEP patients treated for 12 weeks with CLZ vs. 3B+ FEP patients treated with FL-APs
Neutropenia | 12 weeks
  To compare rates of neutropenia in 3B+ FEP patients treated for 12 weeks with CLZ vs. 3B+ FEP patients treated with FL-APs

OTHER OUTCOMES:
Functional MRI | 12 weeks
  Evaluate changes in resting-state functional connectivity patterns related to CLZ response by comparing baseline to 12-week rs-fMRI scans
Functional Outcome | 12 weeks
  To explore the days in hospital of CLZ-treated 3B+ FEP patients vs. 3B+ FEP patients treated with FL-
Functional Outcome | 12 weeks
  To explore suicidal ideation of CLZ-treated 3B+ FEP patients vs. 3B+ FEP patients treated with FL-APs as measured by the CSSRS

CONTACTS AND LOCATIONS:
Locations (1):
- Feinstein Institute for Medical Research, Glen Oaks, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data will be placed in the NDA.
Time Frame: The data will be transferred 12 months after the study starts and then every 6 months
Access Criteria: Access to the NDA will be controlled by the NDA following their policies and procedures.